CLINICAL TRIAL: NCT04901546
Title: Esophageal Atresia: a Natural Experiment of the Effects of Oral Inoculation on the Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, David A. Relman, Professor, Medicine - Infectious Disease, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 58102
Record Dates: First submitted 2021-04-21; First posted 2021-05-25 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Atresia
MeSH Terms: conditions — Esophageal Atresia

STUDY DESIGN:
Intervention Model Description: Infants with esophageal atresia (EA) and comparison infants without esophageal atresia (but also in the neonatal intensive care unit, NICU) will be recruited. Infants with EA will be given their own saliva for 1 week, with every feed. Infants without EA will receive usual care. All subjects will have samples collected according to the same schedule.
  Mothers of infants will also be recruited and have samples collected in order to understand the sources of the infant's gut microbiome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infants with Esophageal Atresia (Experimental): Starting at 3 weeks, infants will be administered 1 mL of their own saliva via gastrostomy tube, with each feed (8x/day) for one week.
  Interventions: Other: Patient's own saliva
- Comparison Infants without Esophageal Atresia (No Intervention): Infants do not have EA and thus can swallow their own saliva.

INTERVENTIONS:
Other: Patient's own saliva — Infants with esophageal atresia will be given their own saliva
  Arms: Infants with Esophageal Atresia

SUMMARY:
The purpose of this study is to understand changes of the gut microbiome due to esophageal atresia. The intervention will be to give a patient his or her own saliva through their gastrostomy tube (directly into the stomach) to observe if this can normalize microbial colonization of the gut.

DETAILED DESCRIPTION:
After being informed about the study and its overall risks, parents will be given the option to enroll their infant. Participants (infants) with esophageal atresia and a gastrostomy tube will be given their own saliva through their gastrostomy tube, directly into the stomach. Samples of saliva and stool will be collected from these infants, and from a comparison group without esophageal atresia, as well as blood and urine to look for changes in immune responses and in metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with Esophageal Atresia (All, no exclusion criteria); maximum age at enrollment is 3 months.
* Neonates matched for gestational age without EA, also anticipated to require surgery (Infants >=32 weeks), or also premature (<32 weeks)

Exclusion Criteria (only for infants without EA):

* sepsis
* admission to study hospital after 7 days old
* expected length of stay <2 weeks

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Change in Gut Microbial Community Structure | From birth until discharge from the hospital, up to 1 year
  Evaluate community structure and differential abundances of dominant taxa and of key taxa to the newborn (e.g., Bifidobacterium, Bacteroides, Lactobacillus, Staphylococcus and Enterobacteriaceae)

SECONDARY OUTCOMES:
Change in Immune System Profile | From birth until discharge from the hospital, up to 1 year
  Determine immune cell profiles using mass cytometry (CyTOF)
Change in Fecal Metabolome Profile | From birth until discharge from the hospital, up to 1 year
  Measure metabolites in the stool using mass spectrometry
Change in Blood Metabolome Profile | From birth until discharge from the hospital, up to 1 year
  Measure metabolites in the blood using mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: David Relman, MD, Principal Investigator — Stanford University; Pearl Houghteling, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No